CLINICAL TRIAL: NCT04488185
Title: An Exploratory, Randomized, Double-blind, Parallel-group, Multicenter Study to Compare Secukinumab 300 mg With Placebo After 16 Weeks of Treatment in Adults With Moderate to Severe Plaque Psoriasis and Subclinical Enthesitis Measured by Musculoskeletal Ultrasound
Brief Title: An Efficacy Study of Secukinumab in Plaque Psoriasis Patients With Subclinical Psoriatic Arthritis as Measured by Musculoskeletal Ultrasound
Acronym: INTERCEPT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457AUS26
Record Dates: First submitted 2020-06-26; First posted 2020-07-27 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Subclinical enthesitis; secukinumab; subclinical psoriatic arthritis; Plaque psoriasis; AIN457
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab 300mg (Experimental): Randomized in a 2:1 ratio to secukinumab or placebo
  Interventions: Biological: Secukinumab 300 mg
- Placebo (Placebo Comparator): Randomized in a 2:1 ratio to secukinumab or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Secukinumab 300 mg — Secukinumab 300 mg administered s.c. (2 single-use prefilled syringes of 150 mg/mL), on Days 1, 8, 15, 22, 29, 57, 85.
  Other Names: AIN457
  Arms: Secukinumab 300mg
Other: Placebo — Placebo administered s.c. (2 single-use prefilled 1 mL syringes) on Days 1, 8, 15, 22, 29, 57, 85.
  Arms: Placebo

SUMMARY:
Given the role of IL-17 in the development of entheseal-driven pathology, a therapeutic strategy aimed at blocking IL-17 would be a logical option for the treatment of subclinical enthesitis in psoriasis patients. This study will be the first randomized trial of a biologic therapy versus placebo in participants with plaque psoriasis and subclinical psoriatic arthritis, using musculoskeletal ultrasound.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the difference in effect between secukinumab 300 mg s.c. and placebo, based on change from baseline to Week 16 in the OMERACT ultrasound enthesitis score.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic plaque-type psoriasis confirmed through physical examination by a dermatologist, with at least six months of clinical history prior to the baseline visit
* Moderate to severe plaque psoriasis at baseline as defined as:
* ≥ 10 % Body Surface Area (BSA) involvement, or
* ≥ 3% to <10% Body Surface Area with involvement of special regions (nails, scalp, or intertriginous skin), or with a history of psoriatic arthritis in a parent

Candidate for systemic therapy, defined as having psoriasis inadequately controlled by current topical and/or systemic treatment(s) (including topical corticosteroids), phototherapy, or previous systemic therapies

Presence of sonographic enthesitis at screening, in at least one enthesis, defined by the presence of at least abnormal thickening and hypoechogenicity of the tendon insertion, with or without presence of Doppler signal (Grade 0-3), or by the presence of grade ≥ 2 Doppler signal, independent of gray scale abnormalities

Exclusion Criteria:

* Diagnosis of PsA as per CASPAR confirmed by a rheumatologist (including the presence of inflammatory pain in entheses or joints), and any other known rheumatological disease affecting the assessed joints
* Exposure to any IL-17 or IL-23(p19) inhibitor for the treatment of psoriasis (approved or investigational) within twelve months prior to screening, or exposure to any inhibitors of TNF-ɑ and IL12/23 within six months prior to screening
* Previous exposure to non-biologic systemic therapy for psoriasis, including methotrexate, PDE-4 inhibitors, or systemic corticosteroids within 12 weeks or 5 half-lives (whichever is longer) prior to screening
* A degree of obesity that impedes proper ultrasound examination of entheses and joints
* Forms of diagnosed psoriasis other than chronic plaque psoriasis (e.g., erythrodermic, generalized or localized pustular psoriasis, or new onset guttate psoriasis)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Outcome Measures in Rheumatology (OMERACT) ultrasound enthesitis score | Baseline and Week 16
  Twelve (12) entheses (bilateral AT, LE, PP, DP, PA, QT) will be scored in terms of inflammatory and morphological components according to the OMERACT enthesitis composite semi-quantitative scale (0 to 3). The lowest OMERACT score a participant can have at baseline is 2 (based on Inclusion Criterion number 6, which requires at least 2 points in the B-mode or the Doppler mode in at least one enthesis). The highest OMERACT score expected at baseline will be 72, assuming that each of the 12 entheses assessed shows a maximum of 3 points in the gray scale score, and a maximum of 3 points in the Doppler score. The largest change expected from baseline to Week 16 is -60 points (improvement). This assumes that the presence of structural changes (calcifications, enthesophytes and erosions) may add a maximum of 12 points to the score, and it may not be modifiable with study treatment during the study period.

SECONDARY OUTCOMES:
Change from Baseline in the Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) ultrasound enthesitis score | Baseline and Week 16
  Sixteen (16) entheses (bilateral AT, LE, PP, DP, PA, QT, SS, TT) will be scored in terms of inflammatory components according with the GRAPPA ultrasound enthesitis score. The lowest GRAPPA score a participant may have at baseline is 2 (based on Inclusion Criterion number 6, which requires at least 2 points in the B-mode or the Doppler mode in at least 1 enthesis). The highest GRAPPA score expected at baseline is 248, assuming the maximum score that could be assigned to each enthesis. The largest change expected from baseline to Week 16 is -136 points (improvement). This value assumes that the presence of structural changes (calcifications, enthesophytes, and erosions) may add a maximum of 136 points to the score, and it may not be modifiable with study treatment during the study period.
Change from Baseline in the PsASon13 unilateral ultrasound composite score of synovitis | Baseline and Week 16
  Joints examined by the PsASon13 unilateral ultrasound composite score: Small finger joints: MCP2, MCP5, H-PIP1, H-PIP2, H-PIP3; Distal interphalangeal finger joints: H-DIP3; Small joints of feet: MTP1, MTP5, F-PIP1; Distal interphalangeal joints of feet: F-DIP2, F-DIP3; Large joints: wrist and knee. Lowest score a participant may have at baseline is 0. Highest score a participant may have at baseline is 184 (5 small finger joints, each ranging from 0 to 18; 1 distal interphalangeal finger joint, each ranging from 0 to 16; 3 small joints of feet, each ranging from 0 to 12; 2 distal interphalangeal joints of feet, each ranging from 0 to 12; 1 wrist ranging from 0 to 12; and 1 knee ranging from 0 to 6). Largest change expected from baseline to Week 16 is -118 points (improvement). This assumes that the presence of structural changes (erosions and osteophytes) may add a maximum of 66 points to the score and it may not be modifiable with study treatment during the study period.
Number of participants who achieve complete resolution of enthesitis based on OMERACT criteria (yes, no) | Baseline and Week 16
  Proportion of participants experiencing complete resolution of their enthesitis based on Change from Baseline in the Outcome Measures in Rheumatology (OMERACT) score
Number of participants who achieve Psoriasis Area and Severity Index 90 (PASI 90) (yes, no) | Baseline and Week 16
  Psoriasis Area Severity Index 90
  Scores range from 0 to 72. A score of more than 10 generally translates to "moderate-to-severe". Usually, the higher your PASI score, the lower the quality of life. A PASI 90 is at least a 90% improvement (reduction) in PASI score.
Number of participants who achieve Psoriasis Area and Severity Index 100 (PASI 100) (yes, no) | Baseline and Week 16
  Psoriasis Area Severity Index 100
  Scores range from 0 to 72. A score of more than 10 generally translates to "moderate-to-severe". Usually, the higher your PASI score, the lower the quality of life. A PASI 100 is a complete clearing of psoriasis (PASI score = 0).
Number of participants who achieve Investigator's Global Assessment modified 2011 (IGA mod 2011) score of 0 or 1 (yes, no) | Baseline and Week 16
  The IGA mod 2011 scale is a visual assessment that consists of a score ranging from 0 (clear) to 4 (severe). Skin rated a 4 is bright red in color with marked plaque elevation and is dominated by thick, non-tenacious scale. For a treatment to be considered successful, the affected area must receive a score of 0 or 1 and experience a two-point improvement from Baseline.
Change from Baseline in Body Surface Area (BSA) | Baseline and Week 16
  The total percentage of body surface area affected by psoriasis
Change from Baseline in Dermatology Life Quality Index (DLQI) score | Baseline and Week 16
  A 10-item measure to assess health-related quality of life in adults with skin diseases. Scores range from 0-30 with a higher score being less quality of life.
Number of participants who achieve Dermatology Life Quality Index (DLQI) score of 0 or 1 (yes, no) | Baseline and Week 16
  A 10-item measure to assess health-related quality of life in adults with skin diseases. Scores range from 0-30 with a higher score being less quality of life.
Change from Baseline in HAQ-DI score | Baseline and Week 16
  Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question scale assessing functional ability. The final HAQ-DI score ranges from 0 (no problems functioning) to 3 (not able to function).
Number of participants who achieve HAQ-DI change from baseline ≤ -0.35 (yes, no) | Baseline and Week 16
  Health Assessment Questionnaire-Disability Index (HAQ-DI) is a 20-question scale assessing functional ability. The final HAQ-DI score ranges from 0 (no problems functioning) to 3 (not able to function).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Acquitter M, Misery L, Saraux A, Bressollette L, Jousse-Joulin S. Detection of subclinical ultrasound enthesopathy and nail disease in patients at risk of psoriatic arthritis. Joint Bone Spine. 2017 Dec;84(6):703-707. doi: 10.1016/j.jbspin.2016.10.005. Epub 2016 Dec 5. PMID 27932277
- [Background] Armstrong AW, Robertson AD, Wu J, Schupp C, Lebwohl MG. Undertreatment, treatment trends, and treatment dissatisfaction among patients with psoriasis and psoriatic arthritis in the United States: findings from the National Psoriasis Foundation surveys, 2003-2011. JAMA Dermatol. 2013 Oct;149(10):1180-5. doi: 10.1001/jamadermatol.2013.5264. PMID 23945732
- [Background] Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008 Nov;159(5):997-1035. doi: 10.1111/j.1365-2133.2008.08832.x. Epub 2008 Sep 15. PMID 18795920
- [Background] Cassell SE, Bieber JD, Rich P, Tutuncu ZN, Lee SJ, Kalunian KC, Wu CW, Kavanaugh A. The modified Nail Psoriasis Severity Index: validation of an instrument to assess psoriatic nail involvement in patients with psoriatic arthritis. J Rheumatol. 2007 Jan;34(1):123-9. PMID 17216680
- [Background] Chen M, Kianifard F. A nonparametric procedure associated with a clinically meaningful efficacy measure. Biostatistics. 2000 Sep;1(3):293-8. doi: 10.1093/biostatistics/1.3.293. PMID 12933510
- [Background] Doherty SD, Van Voorhees A, Lebwohl MG, Korman NJ, Young MS, Hsu S, National Psoriasis Foundation. National Psoriasis Foundation consensus statement on screening for latent tuberculosis infection in patients with psoriasis treated with systemic and biologic agents. J Am Acad Dermatol. 2008 Aug;59(2):209-17. doi: 10.1016/j.jaad.2008.03.023. Epub 2008 May 15. PMID 18485527
- [Background] El Miedany Y, El Gaafary M, Youssef S, Ahmed I, Nasr A. Tailored approach to early psoriatic arthritis patients: clinical and ultrasonographic predictors for structural joint damage. Clin Rheumatol. 2015 Feb;34(2):307-13. doi: 10.1007/s10067-014-2630-2. Epub 2014 May 3. PMID 24794490
- [Background] Elnady B, El Shaarawy NK, Dawoud NM, Elkhouly T, Desouky DE, ElShafey EN, El Husseiny MS, Rasker JJ. Subclinical synovitis and enthesitis in psoriasis patients and controls by ultrasonography in Saudi Arabia; incidence of psoriatic arthritis during two years. Clin Rheumatol. 2019 Jun;38(6):1627-1635. doi: 10.1007/s10067-019-04445-0. Epub 2019 Feb 12. PMID 30756253
- [Background] Faustini F, Simon D, Oliveira I, Kleyer A, Haschka J, Englbrecht M, Cavalcante AR, Kraus S, Tabosa TP, Figueiredo C, Hueber AJ, Kocijan R, Cavallaro A, Schett G, Sticherling M, Rech J. Subclinical joint inflammation in patients with psoriasis without concomitant psoriatic arthritis: a cross-sectional and longitudinal analysis. Ann Rheum Dis. 2016 Dec;75(12):2068-2074. doi: 10.1136/annrheumdis-2015-208821. Epub 2016 Feb 25. PMID 26916344
- [Background] Feldman SR, Zhao Y, Shi L, Tran MH. Economic and Comorbidity Burden Among Patients with Moderate-to-Severe Psoriasis. J Manag Care Spec Pharm. 2015 Oct;21(10):874-88. doi: 10.18553/jmcp.2015.21.10.874. PMID 26402388
- [Background] Ficjan A, Husic R, Gretler J, Lackner A, Graninger WB, Gutierrez M, Duftner C, Hermann J, Dejaco C. Ultrasound composite scores for the assessment of inflammatory and structural pathologies in Psoriatic Arthritis (PsASon-Score). Arthritis Res Ther. 2014 Oct 31;16(5):476. doi: 10.1186/s13075-014-0476-2. PMID 25361855
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Background] Gladman DD, Antoni C, Mease P, Clegg DO, Nash P. Psoriatic arthritis: epidemiology, clinical features, course, and outcome. Ann Rheum Dis. 2005 Mar;64 Suppl 2(Suppl 2):ii14-7. doi: 10.1136/ard.2004.032482. PMID 15708927
- [Background] Gottlieb AB, Griffiths CE, Ho VC, Lahfa M, Mrowietz U, Murrell DF, Ortonne JP, Todd G, Cherill R, Marks I, Emady-Azar S, Paul CF; Multi-Centre Investigator Group. Oral pimecrolimus in the treatment of moderate to severe chronic plaque-type psoriasis: a double-blind, multicentre, randomized, dose-finding trial. Br J Dermatol. 2005 Jun;152(6):1219-27. doi: 10.1111/j.1365-2133.2005.06661.x. PMID 15948985
- [Background] Gutierrez M, Filippucci E, De Angelis R, Salaffi F, Filosa G, Ruta S, Bertolazzi C, Grassi W. Subclinical entheseal involvement in patients with psoriasis: an ultrasound study. Semin Arthritis Rheum. 2011 Apr;40(5):407-12. doi: 10.1016/j.semarthrit.2010.05.009. Epub 2010 Aug 5. PMID 20688358
- [Background] Kampylafka E, d'Oliveira I, Linz C, Lerchen V, Stemmler F, Simon D, Englbrecht M, Sticherling M, Rech J, Kleyer A, Schett G, Hueber AJ. Resolution of synovitis and arrest of catabolic and anabolic bone changes in patients with psoriatic arthritis by IL-17A blockade with secukinumab: results from the prospective PSARTROS study. Arthritis Res Ther. 2018 Jul 27;20(1):153. doi: 10.1186/s13075-018-1653-5. PMID 30053825
- [Background] King MT, Fayers PM. Making quality-of-life results more meaningful for clinicians. Lancet. 2008 Mar 1;371(9614):709-10. doi: 10.1016/S0140-6736(08)60324-4. No abstract available. PMID 18313491
- [Background] Manuel O, Kumar D. QuantiFERON-TB Gold assay for the diagnosis of latent tuberculosis infection. Expert Rev Mol Diagn. 2008 May;8(3):247-56. doi: 10.1586/14737159.8.3.247. PMID 18598104
- [Background] Mathew AJ, Bird P, Gupta A, George R, Danda D. Magnetic resonance imaging (MRI) of feet demonstrates subclinical inflammatory joint disease in cutaneous psoriasis patients without clinical arthritis. Clin Rheumatol. 2018 Feb;37(2):383-388. doi: 10.1007/s10067-017-3895-z. Epub 2017 Dec 4. PMID 29204762
- [Background] Naredo E, Moller I, de Miguel E, Batlle-Gualda E, Acebes C, Brito E, Mayordomo L, Moragues C, Uson J, de Agustin JJ, Martinez A, Rejon E, Rodriguez A, Dauden E; Ultrasound School of the Spanish Society of Rheumatology and Spanish ECO-APs Group. High prevalence of ultrasonographic synovitis and enthesopathy in patients with psoriasis without psoriatic arthritis: a prospective case-control study. Rheumatology (Oxford). 2011 Oct;50(10):1838-48. doi: 10.1093/rheumatology/ker078. Epub 2011 Jun 23. PMID 21700682
- [Background] Savage L, Goodfield M, Horton L, Watad A, Hensor E, Emery P, Wakefield R, Wittmann M, McGonagle D. Regression of Peripheral Subclinical Enthesopathy in Therapy-Naive Patients Treated With Ustekinumab for Moderate-to-Severe Chronic Plaque Psoriasis: A Fifty-Two-Week, Prospective, Open-Label Feasibility Study. Arthritis Rheumatol. 2019 Apr;71(4):626-631. doi: 10.1002/art.40778. Epub 2019 Mar 4. PMID 30468001
- [Background] Scher JU, Ogdie A, Merola JF, Ritchlin C. Preventing psoriatic arthritis: focusing on patients with psoriasis at increased risk of transition. Nat Rev Rheumatol. 2019 Mar;15(3):153-166. doi: 10.1038/s41584-019-0175-0. PMID 30742092
- [Background] Tinazzi I, McGonagle D, Biasi D, Confente S, Caimmi C, Girolomoni G, Gisondi P. Preliminary evidence that subclinical enthesopathy may predict psoriatic arthritis in patients with psoriasis. J Rheumatol. 2011 Dec;38(12):2691-2. doi: 10.3899/jrheum.110505. No abstract available. PMID 22134799
- [Background] Villani AP, Rouzaud M, Sevrain M, Barnetche T, Paul C, Richard MA, Beylot-Barry M, Misery L, Joly P, Le Maitre M, Aractingi S, Aubin F, Cantagrel A, Ortonne JP, Jullien D. Prevalence of undiagnosed psoriatic arthritis among psoriasis patients: Systematic review and meta-analysis. J Am Acad Dermatol. 2015 Aug;73(2):242-8. doi: 10.1016/j.jaad.2015.05.001. Epub 2015 Jun 6. PMID 26054432
- [Background] Weisman S, Pollack CR, Gottschalk RW. Psoriasis disease severity measures: comparing efficacy of treatments for severe psoriasis. J Dermatolog Treat. 2003 Sep;14(3):158-65. doi: 10.1080/09546630310013360. PMID 14522626
- [Background] Zabotti A, McGonagle DG, Giovannini I, Errichetti E, Zuliani F, Zanetti A, Tinazzi I, De Lucia O, Batticciotto A, Idolazzi L, Sakellariou G, Zandonella Callegher S, Sacco S, Quartuccio L, Iagnocco A, De Vita S. Transition phase towards psoriatic arthritis: clinical and ultrasonographic characterisation of psoriatic arthralgia. RMD Open. 2019 Oct 23;5(2):e001067. doi: 10.1136/rmdopen-2019-001067. eCollection 2019. PMID 31749987
- [Result] Acquacalda E, Albert C, Montaudie H, Fontas E, Danre A, Roux CH, Breuil V, Lacour JP, Passeron T, Ziegler LE. Ultrasound study of entheses in psoriasis patients with or without musculoskeletal symptoms: A prospective study. Joint Bone Spine. 2015 Jul;82(4):267-71. doi: 10.1016/j.jbspin.2015.01.016. Epub 2015 Apr 13. PMID 25881759